CLINICAL TRIAL: NCT06411340
Title: An Observational-based Registry of Routinely Collected Clinical Parameters to Study Inflammation in Acute Cardiovascular Diseases - the CArdiovascular Inflammation Registry
Brief Title: Inflammation in Acute Cardiovascular Diseases - the CArdiovascular Inflammation Registry (CAIR)
Acronym: CAIR
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 334636
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Inflammation; Cardiovascular Diseases; Myocarditis; Pericarditis; Myocardial Infarction; Heart Failure; Heart Diseases
Keywords: Inflammation; Acute cardiovascular disease; Myocarditis; Registry; Electronic health records; Pericarditis; Myocardial infarction
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases; Myocarditis; Pericarditis; Myocardial Infarction; Heart Failure; Heart Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute inflammatory cardiac disease: This registry aims to collate routinely collected clinical data on patients with acute cardiovascular diseases.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
Following acute cardiovascular injury, inflammation is vital to activate reparative mechanisms. However, there is compelling evidence implicating excessive inflammation and dysregulated resolution in fibrosis, ventricular remodelling, and heart failure (HF). Recently, the anti-inflammatory agent colchicine reduced cardiovascular events after myocardial infarction (MI) compared to placebo, indicating that targeting inflammation in acute cardiovascular conditions is feasible. Several acute cardiovascular conditions are characterised by inflammation, including myocarditis, MI, and acute heart failure. However, there is large variability in definition, epidemiology, clinical presentation, pathophysiology, and natural history of acute inflammatory cardiovascular diseases. This relates, in part, to the difficulty in performing adequately powered studies. Clinical studies that include sufficient patients and extended observation periods are necessary to address some of these knowledge gaps. This registry aims to collate routinely collected clinical data on patients with acute cardiovascular diseases characterised by inflammation in an observational-based registry. By doing so, the investigators hope to understand the contribution of inflammation to the pathophysiology of acute cardiovascular disease, improve risk stratification, and identify potential novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 13 years of age or older with an acute cardiovascular condition requiring hospital admission is eligible.

Exclusion Criteria:

* <13 years of age

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed with acute cardiovascular diseases can be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2034-07 (Estimated); Study Completion 2039-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year
  Primary outcome will include all-cause mortality, but will vary by specific research project conducted within the registry.

IPD SHARING:
Plan to Share IPD: No
Partner sites (including those outside the UK) will store linkage files for their own patients in accordance with local policies. Data will be stored on a research database (REDCap) hosted by King's College London. Each participating centre will have linkage codes for their own patients only. Therefore, exported data will not be identifiable to other centres.